CLINICAL TRIAL: NCT06800820
Title: Determination of Biological Activity of Human-enriched Serum Following Chondractiv™ Plus Ingredient Ingestion : Result From an Exploratory Clinical Trial
Brief Title: Determination of Biological Activity of Human-enriched Serum Following Chondractiv™ Plus Ingredient Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symrise Group (Industry)
Collaborators: Clinic'n'Cell (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CnC2024 - ChondractivPlus
Record Dates: First submitted 2025-01-09; First posted 2025-01-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Collagen hydrolysate

STUDY DESIGN:
Intervention Model Description: Phase 1: 15 healthy volunteers divided in 3 groups
  * Group 1: 5 volunteers taking 1 oral dose of Chondractiv™ Plus 1,5g
  * Group 2: 5 volunteers taking 1 oral dose of Chondractiv™ Plus 4,5g
  * Group 3: 5 volunteers taking 1 oral dose of Chondractiv™ Plus 15g
  Phase 2: 10 volunteers taking 1 dose of Chondractiv™ Plus 15g.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chondractiv™ Plus (Other): Phase 1: One dose of 1,5g or 4,5g or 15g
  Phase 2: One dose of 15g
  Interventions: Dietary Supplement: Chondractiv™ Plus (Hydrolyzed chicken cartilage)

INTERVENTIONS:
Dietary Supplement: Chondractiv™ Plus (Hydrolyzed chicken cartilage) — One oral dose

SUMMARY:
The main objective of this study is, after collecting serum enriched with metabolites of interest resulting from the ingestion of the Chondractiv™ Plus food supplement (an hydrolyzed chicken collagen), to determine the influence of these sera enriched with circulating metabolites on the behavior of human joint cartilage cells placed in culture.

DETAILED DESCRIPTION:
The clinical study will be conducted in two phases.

1. The first phase will aim at characterizing the metabolites present in human serum after consumption of the Chondractiv™ ingredient and at determining the overall absorption peak of the tested ingredient.
2. The second phase will involve collecting sera enriched with metabolites at the absorption peak, following the ingestion of the ingredient. Subsequently, the final objective will be to characterize the influence of these sera enriched with metabolites of interest on the behavior of human joint cartilage cell cultures.

ELIGIBILITY:
Inclusion Criteria:

* Liver function tests within reference norms.
* Kidney function tests within reference norms.
* Complete blood count (CBC) within reference norms.
* C-reactive protein (CRP) within reference norms.
* Blood pressure compatible with study requirements.
* Non-smoker or occasional smoker (max 5 cigarettes/day or max 10 ml per week of e-liquid with a nicotine concentration of 3 mg/ml).
* Maximum 5 hours of intense sports per week.
* Weight ≥ 60 kg.
* Body Mass Index (BMI) between 20 and 28 kg/m² (exclusive).
* Subjects who are able and willing to comply with the protocol and give their informed written consent.
* Subjects affiliated with the social security.

Exclusion Criteria:

* Any type of vaccination within the past month.
* Alcohol consumption exceeding WHO standards (Sup. 3 drinks per day for men).
* Ongoing treatment (medication, dietary supplement, or probiotic) and within the four weeks prior to inclusion.
* Known pathology (including seasonal).
* Allergy to the study product
* Individuals following a diet unsuitable for the study (e.g., vegetarian, vegan, or plant-based diets).
* Change in eating habits within the 4 weeks prior to inclusion.
* Medical and/or surgical history deemed incompatible with the trial by the investigator or their representative.
* Persons under guardianship, curatorship, deprived of freedoms, safeguarding justice.
* Refusal to sign the information sheet and consent

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Biological activity of human-enriched serum following Chondractiv™ Plus ingredient ingestion | T0 and Tmax (within 180 minutes after Chondractiv™ Plus ingredient ingestion, time determined during phase 1 described in secondary outcome)
  The main objective of this study is to determine the influence of human serum enriched with metabolites from ingestion of Chondractiv™ Plus on the behavior of human primary chondrocyte cultures (phase 2).

SECONDARY OUTCOMES:
Concentration of circulating amino-acids including hydroxyproline in blood stream. The aim is to characterize the absorption kinetics profile of Chondractiv™ Plus according to the dose ingested (phase 1). | From blood draw at different time points (T0, T30, T60, T90, T120, T180 minutes) over the 3 hours following the ingestion of the Chondractiv™ Plus
  Characterize the absorption kinetics profile of Chondractiv™ Plus according to the dose ingested by measuring the circulating metabolites level and in particular amino acids such as hydroxyproline - present in the ingredient (phase 1).
Proteomic | From blood draw at different time points (T0, T30, T60, T90, T120, T180 minutes) over the 3 hours following the ingestion of the Chondractiv™ Plus
  Characterize changes in plasma proteome after consumption of the ingredient Chondractiv™ Plus (phase 1).

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, PhD, Principal Investigator — CIC Clermont-Ferrand
Locations (1):
- Centre d'Investigation Clinique (PIC/CIC), Bâtiment 3C - 58, rue Montalembert, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No